CLINICAL TRIAL: NCT06813781
Title: A Phase I, Multicentre, Single-Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD5004
Brief Title: Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD5004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea Clinical Research Unit Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7260C00011
Record Dates: First submitted 2024-12-17; First posted 2025-02-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Healthy participants; AZD5004; Pharmacokinetics; Safety

STUDY DESIGN:
Intervention Model Description: Up to four groups (three hepatic impairment groups and controls with normal hepatic function) will be enrolled into this study.
  All participants will receive the study intervention:
  * Cohort 1 will enroll 8 participants with mild hepatic impairment
  * Cohort 2 will enroll 8 participants with moderate hepatic impairment
  * Cohort 3 will enroll 6-8 participants with severe hepatic impairment
  * Cohort 4 will enroll ~8 participants with normal hepatic function matched by sex, age, and body weight
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): A single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004
- Group 2 (Experimental): A single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004
- Group 3 (Experimental): A single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004
- Group 4 (Experimental): A single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004

INTERVENTIONS:
Drug: AZD5004 — Dose 1
  Other Names: ECC5004; Dose 1

SUMMARY:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD5004 in male and female participants with mild, moderate, and severe hepatic impairment compared with participants with normal hepatic function.

DETAILED DESCRIPTION:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD5004 in male and female participants with mild, moderate, or severe hepatic impairment compared with participants with normal hepatic function.

Participants will be enrolled within the following groups based on their Child Pugh classification score as determined at screening:

Group 1: Participants with mild hepatic impairment (Child Pugh Class A, score of 5 or 6).

Group 2: Participants with moderate hepatic impairment (Child Pugh Class B, score of 7 to 9).

Group 3: Participants with severe hepatic impairment (Child Pugh Class C, score of 10 to 15).

Group 4: Participants with normal hepatic function matched on a group level regarding sex, age, and body weight to the impaired participants.

ELIGIBILITY:
Inclusion Criteria:

For ALL participants:

* Adults 18-80 years of age
* Weight ≥50kg and BMI between ≥18 to ≤40 kg/m2 For participants with normal hepatic function:
* Participant must be stable on a concomitant medication and/or treatment regimen for at least 2 weeks prior to screening

For Healthy Controls:

-Participant must be medically healthy with no significant findings on medical evaluation at screening to include but not limited to an eGFR >90 ml/min/1.73 m2

For participants with hepatic impairment:

* Group 1 (mild) must have an Child-Pugh score of 5 or 6, Group 2 (moderate) must have a Child-Pugh score of 7 to 9, Group 3 (severe) must have a Child-Pugh score of 10 to 15.
* Participant must have a diagnosis of chronic (≥ 6 months) and stable hepatic impairment (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status within 30 days prior to study screening

Exclusion Criteria:

For ALL participants:

* Poorly controlled diabetes mellitus (A1C >10% at screening).
* Unwillingness to use adequate contraception
* Uncontrolled hypertension or hypotension
* Presence of unstable systemic disease or psychologic conditions.
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG.

Specific For Healthy Controls:

-Positive screening for HIV, Hepatitis B, or Hepatitis C -

-Any clinically significant disease or disorder to include but not limited to acute or chronic liver disease

Specific For Hepatically Impaired Participants:

* eGFR <60 ml/min/1.73 m2
* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment to include rising LFTs, paracentesis at less than 4 week intervals, oesophageal banding within the last 3 months, or treatment for GI bleeding within the last 6 months
* Presence of a hepatocellular carcinoma or acute liver disease caused by an infection or drug toxicity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
AUCinf | Day 1 to Day 6
  Area under plasma concentration-time curve from zero to infinity
AUClast | Day 1 to Day 6
  Area under plasma concentration-time curve from time zero to the last measurable concentration
Cmax | Day 1 to Day 6
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Tmax | Day 1 to Day 6
  Time to reach maximum observed plasma concentration
PK parameters (t1/2λz) | Day 1 to Day 6
  Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve
PK parameters CL/F | Day 1 to Day 6
  Apparent total body clearance of drug from plasma after extravascular administration
PK parameters CLNR/F | Day 1 to Day 6
  Non-renal clearance of drug from plasma after oral administration
PK parameter Vz/F | Day 1 to Day 6
  Apparent volume of distribution during the terminal phase after extravascular administration
PK parameter CLr | Day 1 to Day 6
  Renal clearance of the drug from plasma
PK parameter Ae | Day 1 to Day 6
  Cumulative amount of unchanged drug excreted into the urine
fe | Day 1 to Day 6
  Fraction of the drug excreted into the urine

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | Day 1 to Day 10
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Participants with abnormal blood pressure | Day 1 to Day 6
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Number of participants with abnormal laboratory tests results | Day 1 to Day 6
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Number of participants with serious adverse events (SAEs) | Day 1 to Day 10
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Participants with abnormal ECG QTcF findings | Day 1 to Day 6
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Participants with abnormal physical examination findings | Day 1 to Day 6
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Participants with abnormal heart rate | Day 1 to Day 6
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function
Number of participants with abnormal ECG PR interval findings | Day 1 to Day 6
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with mild, moderate, and severe hepatic impairment and those with normal hepatic function

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Lake Forest, California
  - Research Site, Rialto, California
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home